CLINICAL TRIAL: NCT00582738
Title: A Randomized, Controlled, Open Label, Two Arms, Exploratory Study to Evaluate the Effect of Everolimus on Histologically Assessed Fibrosis Progression (Ishak-Knodell) in Liver Transplant Recipients With Recurrent Hepatitis C Viral Infection as Compared to Standard Treatment.
Brief Title: Efficacy of Everolimus as Inhibitor of Fibrosis Progression in Liver Transplant Patients With Recurrence of Hepatitis C Viral Infection
Acronym: REVERT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001H2301
Record Dates: First submitted 2007-12-12; First posted 2007-12-28 (Estimated); Results first posted 2012-09-06 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-08

CONDITIONS: Recurrent Hepatitis C
Keywords: Fibrosis progression; recurrent hepatitis C; viral infection; liver transplant recipients; everolimus; Hepatitis C recurrence after orthotopic liver transplantation (OLT)
MeSH Terms: conditions — Hepatitis C; Virus Diseases | interventions — Everolimus

ARMS (2):
- CsA-TAC (Active Comparator): Continuation of current immunosuppressive regimen (continuation of Calcineurin Inhibitor [CNI] with or without Enteric-coated mycophenolate sodium (myfortic) or mycophenolate mofetil(Cellcept)[MPA], with or without steroids) / no everolimus introduction.
  Interventions: Drug: CsA-TAC (standard Treatment)
- everolimus (Experimental): Initiation of everolimus with discontinuation of CNI/MPA, with or without steroids.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: CsA-TAC (standard Treatment) — Continuation of current immunosuppressive regimen (continuation of CNI with or without MPA, with or without steroids) / no everolimus introduction.
  Arms: CsA-TAC
Drug: Everolimus — Hepatitis C recurrence after orthotopic liver transplantation (OLT)
  Arms: everolimus

SUMMARY:
This study will assess the efficacy of everolimus as an inhibitor of fibrosis progression in liver transplant patients who have a recurrence of hepatitis C viral infection in the transplant

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 - 65 years of age
* Recipients of deceased or living donors
* Patients who had undergone primary liver transplantation at least 6 months before enrolment
* Recurrent Hepatitis C viral infection and histologically confirmed liver fibrosis (stage I-IV in the Ishak-Knodell scale) obtained at baseline or within the previous 6 months to the date of enrolment
* Patients receiving tacrolimus or cyclosporine micro-emulsion with or without - Mycophenolic acid (MPA), with or without steroids.
* Absence of acute rejection episodes within the previous 6 months to the date of enrolment
* Patient in whom an allograft biopsy will not be contraindicated
* Patient willing and capable of giving written informed consent for study participation and able to participate in the study for 24 months
* Patients with Hepatocellular carcinoma (HCC) within the University California, San Francisco (UCSF) Criteria and no recurrence for at least 18 months after OLT.

Exclusion Criteria:

* Recipients of multiple organ transplants or patients who have undergone retransplantation
* Current biliary complications
* History of drug or alcohol abuse within 1 year before enrolment
* Patients treated with anti-hepatitis C virus treatment at the time of enrollment or within the previous month to the date of enrolment
* Co-infection with Hepatitis B virus (HBV) or Human Immunodeficiency Virus (HIV)
* Patients with Leukocyte count (WBC) < 3000/mm3, platelet count < 75000/mm3 or Hemoglobin (Hb) < 8 g/dl
* Patients with proteinuria >1g/24 hours
* Patient with a current severe systemic infection

Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative site, Buenos Aires, Argentina

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Treatment: Continuation of current immunosuppressive regimen (continuation of Calcineurin Inhibitor [CNI] with or without Enteric-coated mycophenolate sodium (myfortic) or mycophenolate mofetil(Cellcept)[MPA], with or without steroids) / no everolimus introduction.
Period: Overall Study
Arm/Group | Standard Treatment | Everolimus
Started | 21 | 22
Completed | 12 | 4
Not Completed | 9 | 18
Not completed — Administrative Problems | 7 | 8
Not completed — Adverse Event | 0 | 5
Not completed — Graft Lost | 0 | 1
Not completed — Other | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment | Everolimus | Total
Number analyzed (Participants) | 21 | 22 | 43
Age Continuous [Median (Full Range); unit: years] | 60.0 (6.79) [43 to 70] | 56.5 (8.01) [41 to 69] | 57 [41 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 11 | 15 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fibrosis Staging Score (Measured by the Ishak-Knodell Staging Score) Between Baseline and 24 Months Post-transplant.
Description: Ishak-Knodell Score: 0=No fibrosis; 01=Fibrous expansion of some portal areas, with or without short fibrous septa; 02=Fibrous expansion of most portal areas, with or without short fibrous septa; 03=Fibrous expansion of most portal areas, with occasional portal to portal (P-P) bridging; 04=Fibrous expansion of portal areas, with marked bridging (portal to portal (P-P) as well as portal to central (P-C)); 05=Marked bridging (P-P and/or P-C) with occasional nodules (incomplete cirrhosis); 06=Cirrhosis, probable or definite
  Decrease in score from baseline indicates improvement
Time Frame: baseline, 24 Months
Population: The Intent to Treat (ITT) population consisted of all patients randomized and who had at least one dose of study medication. Small number of biopsies obtained at Month 24 due to study being prematurely terminated.
Measure: Median (Full Range); unit: Score on Scale
Arm/Group | CsA-TAC | Everolimus
Number analyzed (Participants) | 8 | 5
Score on Scale | -0.5 (1.20) [-1.0 to 2.0] | 0.0 (0.45) [-1.0 to 0.0]

2. Secondary Outcome: Change From Baseline in Fibrosis Metavir Scoring at 12 and 24 Months Post Randomization
Description: Metavir Score: F0=No fibrosis; F1=Portal fibrosis without septa; F2=Portal fibrosis with rare septa; F3=Numerous septa without cirrhosis Decrease in score from baseline indicates improvement
Time Frame: Baseline, 12 months, 24 months
Population: The Intent to Treat (ITT) population consisted of all patients randomized and who had at least one dose of study medication. Only participants with observations at baseline and specified timepoints were included in the analysis.
Measure: Median (Full Range); unit: Scores on a Scale
Arm/Group | CsA-TAC | Everolimus
Number analyzed (Participants) | 18 | 14
Scores on a Scale
  Baseline (n=18, 14) | 1.0 (0.84) [1.0 to 4.0] | 1.5 (0.83) [1.0 to 3.0]
  Month 12 (n=18, 14) | 1.0 (1.04) [0.0 to 4.0] | 1.0 (0.80) [0.0 to 3.0]
  Month 24 (n=8, 5) | 1.0 (1.04) [0.0 to 3.0] | 1.0 (0.89) [1.0 to 3.0]
  Month 12-Baseline (n=18, 14) | 0.0 (0.76) [-1.0 to 2.0] | 0.0 (0.85) [-2.0 to 1.0]
  Month 24-Baseline (n=8, 5) | 0.0 [-1.0 to 2.0] | 0.0 [-1.0 to 0.0]

3. Secondary Outcome: Percentage of Patients With Death, Graft Loss and Biopsy Proven Acute Rejection (BPAR) Between Study Groups
Time Frame: 24 Months
Population: The Intent to Treat (ITT) population consisted of all patients randomized and who had at least one dose of study medication.
Measure: Number; unit: Percentage of Participants
Groups:
- CsA/TAC: Continuation of current immunosuppressive regimen (continuation of Calcineurin Inhibitor [CNI] with or without Enteric-coated mycophenolate sodium (myfortic) or mycophenolate mofetil(Cellcept)[MPA], with or without steroids) / no everolimus introduction.
Arm/Group | CsA/TAC | Everolimus
Number analyzed (Participants) | 21 | 22
Percentage of Participants
  Death | 0 | 4.5
  Graft Loss | 0 | 4.5
  Acute Rejection (BPAR) | 0 | 0.0

4. Secondary Outcome: Number of Patients With Events (Progression to Cirrhosis, Retransplantation, HCV Related Death, First BPAR, Graft Loss)at 12 and 24 Months
Time Frame: 12 months, 24 months
Population: The Intent to Treat (ITT) population consisted of all patients randomized and who had at least one dose of study medication. During different time points, participants with observations at that time point were included in the analysis.
Measure: Number; unit: participants
Arm/Group | CsA-TAC | Everolimus
Number analyzed (Participants) | 21 | 22
participants
  12 months | 0 | 0
  24 months | 0 | 1

5. Secondary Outcome: Comparison of Renal Function (Glomerular Filtration Rate [GFR] Calculated Using the Modification of Diet in Renal Disease Study Group [MDRD] Formula) Between Study Groups
Description: GFR Month 9 value if available, otherwise minimal first year post-randomization available value. Imputation rule of missing Month 24 GFR values: GFR Month 18 value if available, otherwise Month 12 GFR is used.
  Least square means are from an ANCOVA model containing treatment as factor and baseline eGFR as a covariate.
Time Frame: 12 months, 24 months/EOS
Population: The Intent to Treat (ITT) population consists of all patients randomized and who have at least one dose of study medication. During different time points, participants with observations at that time point were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73^2
Arm/Group | CsA-TAC | Everolimus
Number analyzed (Participants) | 21 | 22
mL/min/1.73^2
  12 Months (n=21, 22) | 62.2 (2.95) | 65.6 (2.88)
  24 months (n=20, 18) | 65.5 (2.51) | 71.6 (2.65)

6. Secondary Outcome: Comparison of the Effect of Both Regimens in the Necroinflammatory Grading Score (Ishak-Knodell) (Portal Inflammation)
Description: Ishak-Knodell Score: 0=No fibrosis; 01=Fibrous expansion of some portal areas, with or without short fibrous septa; 02=Fibrous expansion of most portal areas, with or without short fibrous septa; 03=Fibrous expansion of most portal areas, with occasional portal to portal (P-P) bridging; 04=Fibrous expansion of portal areas, with marked bridging (portal to portal (P-P) as well as portal to central (P-C)); 05=Marked bridging (P-P and/or P-C) with occasional nodules (incomplete cirrhosis); 06=Cirrhosis, probable or definite
Time Frame: baseline, 12 months, 24 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | CsA-TAC | Everolimus
Number analyzed (Participants) | 18 | 14
Score on a scale
  Baseline (n= 18, 14) | 1.8 (1.04) | 2.4 (.93)
  Month 12 (n = 18, 14) | 1.9 (1.02) | 1.9 (1.00)
  Month 24 (n = 8, 5) | 2.1 (0.35) | 2.0 (0.71)

7. Secondary Outcome: Comparison of the Effect of Both Regimens on the Inflammatory (Acti-test) and Fibrosis (Fibro-test) Components of Fibrosure, and on Fibrosis Area Assessed by Histomorphometry
Description: The Fibrosure test is the combination of Fibro-test + Acti-test.
  FibroTest (FT) was for the assessment of fibrosis. Fibro test was calculated using an original combination of five highly concentrated serum biochemical markers; alpha2macroglobulin, haptoglobin, apolipoprotein A1, total bilirubin and gammaglutamyltransferase (GGT). FibroTest scores range from 0.00 to 1.00 where 0.0-0.21 is no fibrosis and >= 0.59 is cirrhosis.
  Acti-test was calculated using 6 serum biochemical markers; alpha2macroglobulin, haptoglobin, apolipoprotein A1, total bilirubin, GGT and alanine aminotransferase (ALT). ActiTest (AT) was used for the assessment of necroinflammatory activity. Test score ranges from 0.00 to 1.00, where 0.00-0.17 indicates no necrosis and >= 0.61 indicates severe necrosis
  If 12-month Actitest value was the last available assessment, the value is used to impute the final staging score(End of Study)
Time Frame: baseline, 12 and 24 months
Population: as for outcome 5
Measure: Median (Full Range); unit: units on a scale
Groups:
- Standard Treatment - Summary of Actitest by Treatment; Standard Treatment -Summary of Fibrotest by Treatment: Continuation of current immunosuppressive regimen (continuation of Calcineurin Inhibitor [CNI] with or without Enteric-coated mycophenolate sodium (myfortic) or mycophenolate mofetil(Cellcept)[MPA], with or without steroids) / no everolimus introduction.
- Everolimus -Summary of Actitest by Treatment; Everolimus - Summary of Fibrotest by Treatment: Initiation of everolimus with discontinuation of CNI/MPA, with or without steroids.
Arm/Group | Standard Treatment - Summary of Actitest by Treatment | Everolimus -Summary of Actitest by Treatment | Standard Treatment -Summary of Fibrotest by Treatment | Everolimus - Summary of Fibrotest by Treatment
Number analyzed (Participants) | 21 | 22 | 21 | 21
units on a scale
  Baseline (n=21,21,21,21) | 0.40 (.30) [0.10 to 0.90] | 0.50 (.25) [0.20 to 1.0] | 0.80 (.18) [0.40 to 1.0] | 0.80 (.13) [0.50 to 1.0]
  month 12 (n=20,17, 20, 17) | 0.60 (.28) [0.0 to 0.90] | 0.50 (.23) [0.20 to 1.0] | 0.80 (.16) [0.40 to 1.0] | 0.80 (.15) [0.40 to 1.0]
  month 24 (n=1,2,1,2) | 0.60 (0.0) [0.60 to 0.60] | 0.70 (.33) [0.40 to 0.90] | 0.90 (0.0) [0.90 to 0.90] | 1.0 (.04) [0.90 to 1.0]
  end of study [month 24] (n=20,21,20,21) | 0.60 (.32) [0.10 to 0.90] | 0.50 (.26) [0.10 to 1.0] | 0.80 (.15) [0.50 to 1.0] | 0.70 (.17) [0.50 to 1.0]

8. Secondary Outcome: Percentage of Patients in Each Study Arm With Increase of ≥1 Point in the Ishak-Knodell Staging Score in Fibrosis
Description: as for outcome 6
Time Frame: baseline to month 24
Population: Difference Ishak-Knodell Score at End-of-Study The Intent to Treat (ITT) population consists of all patients randomized and who have at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Standard Treatment | Everolimus
Number analyzed (Participants) | 21 | 22
percentage of participants | 38.9 | 7.1

9. Secondary Outcome: Change From Baseline in Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Viral Load at 12 and 24 Months Post Randomization
Description: End of Study (EOS) endpoint is the last available assessment on or after Month 12. A reduction of at least two logs in HCV RNA viral load was considered as success
Time Frame: baseline, 12 months, 24 months/EOS
Population: The Intent to Treat (ITT) population consists of all patients randomized and who have at least one dose of study medication. If 12-month HCV was the last available assessment, this value is used to impute the End of Study value.
Measure: Mean (Standard Deviation); unit: log10 copies/ml
Arm/Group | CsA-TAC | Everolimus
Number analyzed (Participants) | 20 | 20
log10 copies/ml
  baseline | 6.6 (0.69) | 6.4 (0.94)
  12 months (n=20, 20) | 6.5 (0.84) | 6.6 (.85)
  24 months/EoS (n=20, 20) | 6.9 (0.69) | 6.7 (0.87)
  Month 12 - baseline (n=20,20) | -0.1 (0.71) | 0.2 (0.72)
  Monh 24 - baseline (n=20,20) | 0.3 (0.76) | 0.3 (0.84)

ADVERSE EVENTS:
Groups:
- CsA/TAC: Continuation of current immunosuppressive regimen (continuation of CNI with or without MPA, with or without steroids) / no everolimus introduction.
- EVR (Everolimus): Initiation of everolimus with discontinuation of CNI/MPA, with or without steroids.
Arm/Group | CsA/TAC | EVR (Everolimus)
Serious Adverse Events (participants affected / at risk) | 0/21 | 11/22
Other Adverse Events (participants affected / at risk) | 8/21 | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CsA/TAC (N=21) | EVR (Everolimus) (N=22)
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Hepatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CsA/TAC (N=21) | EVR (Everolimus) (N=22)
Leukopenia (Blood and lymphatic system disorders) | 1 | 2
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Mouth ulceration (Gastrointestinal disorders) | 1 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 3
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Bronchitis (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Blood cholesterol increased (Investigations) | 2 | 3
Blood triglycerides increased (Investigations) | 2 | 1
Blood uric acid abnormal (Investigations) | 2 | 0
Blood uric acid increased (Investigations) | 2 | 0
Liver function test abnormal (Investigations) | 0 | 4
Platelet count decreased (Investigations) | 0 | 3
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 3
Proteinuria (Renal and urinary disorders) | 2 | 2
Renal impairment (Renal and urinary disorders) | 4 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 5
Hypertension (Vascular disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.